CLINICAL TRIAL: NCT05913635
Title: Effects of Time-Restricted Fasting on the Postprandial Glycemic Responses in Chinese Adults: A Randomized Crossover Study
Brief Title: Effects of Time-Restricted Fasting on the Postprandial Glycemic Responses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yuwei Liu, Associate Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 21PJD005
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Time-Restricted Fasting; Postprandial Blood Glucose; Continuous Glucose Monitoring; Crossover trial
MeSH Terms: conditions — Intermittent Fasting | interventions — Lunch; Meals; Breakfast

STUDY DESIGN:
Intervention Model Description: A randomized, crossover study design uses two intervention days (a no-breakfast day and a no-dinner day) and a 6-day washout period.
Who Masked: Outcomes Assessor
Masking Description: The researchers who conducted the biomarker measurements were not aware of the assignments of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-breakfast (Experimental): One-day meal plan with no breakfast. The dietary plan has been developed according to the Dietary Guidelines for Chinese Residents (2022), and the energy distribution of the two meals (lunch and dinner) is 1:1, with the energy percentage of carbohydrates, proteins, and fats being 55%, 15%, and 30%, respectively. The total daily calorie intake has been calculated based on the gender difference of the participants. Since the recommended daily calorie intake for males is 2000 kcal while for females it is 1600 kcal, each meal for males is designed to provide 667 kcal calories, comprising 92g carbohydrates, 22g fat, and 25g protein; each meal for females is designed to provide 533 kcal calories, comprising 73g carbohydrates, 18g fat, and 20g protein. The carbohydrates are sourced from buckwheat flour and mixed grain rice, which create similar glycemic indexes for each meal. Additionally, the one-day meal for both males and females includes 450g of vegetables and 320g of fruits.
  Interventions: Behavioral: Consumption of lunch and dinner, with no breakfast
- No-dinner (Experimental): One-day meal plan with no dinner. The dietary plan has been developed according to the Dietary Guidelines for Chinese Residents (2022), and the energy distribution of the two meals (breakfast and lunch) is 1:1, with the energy percentage of carbohydrates, proteins, and fats being 55%, 15%, and 30%, respectively. The total daily calorie intake has been calculated based on the gender difference of the participants. Since the recommended daily calorie intake for males is 2000 kcal while for females it is 1600 kcal, each meal for males is designed to provide 667 kcal calories, comprising 92g carbohydrates, 22g fat, and 25g protein; each meal for females is designed to provide 533 kcal calories, comprising 73g carbohydrates, 18g fat, and 20g protein. The carbohydrates are sourced from buckwheat flour and mixed grain rice, which create similar glycemic indexes for each meal. Additionally, the one-day meal for both males and females includes 450g of vegetables and 320g of fruits.
  Interventions: Behavioral: Consumption of breakfast and lunch, with no dinner

INTERVENTIONS:
Behavioral: Consumption of lunch and dinner, with no breakfast — The day before intervention day, all participants will be provided with 3 nutritionally balanced meals which are designed by the investigators. On the no-breakfast intervention day, participants are instructed to fast and only be allowed to consume water until 1.00 p.m. and consume the above-designed lunch and dinner at 1.00 p.m. and 8.00 p.m. Additionally, all participants are informed that they are only allowed to consume water between meals and before receiving breakfast at 7.30 a.m. the following day.
  Arms: No-breakfast
Behavioral: Consumption of breakfast and lunch, with no dinner — The day before intervention day, all participants will be provided with 3 nutritionally balanced meals which are designed by the investigators. On the no-dinner intervention day, participants are instructed to consume the above-designed breakfast and lunch at 7.30 a.m. and 1.00 p.m., and no dinner. Additionally, all participants are informed that they are only allowed to consume water between meals and before receiving breakfast at 7.30 a.m. on the following day.
  Arms: No-dinner

SUMMARY:
The goal of this clinical trial is to investigate whether fasting timing has a significant effect on postprandial glycemic responses in healthy adults. The main questions it aims to answer are:

1. Whether fasting timing has a significant effect on postprandial insulin actions and plasma glucose concentration.
2. Whether fasting timing could modulate the glycemic metabolome and circadian rhythms in healthy individuals.

Participants will get the two interventions:

No-dinner: breakfast at 7.30 a.m., lunch at 1.00 p.m. and no dinner; No-breakfast: no breakfast, lunch at 1.00 p.m. and dinner at 8.00 p.m.

DETAILED DESCRIPTION:
A randomized, crossover study design is used with 2 intervention days and a 6-day washout period, to evaluate the effects of early and late fasting on postprandial glucose responses in healthy adults. Randomization was performed by the Fudan staff with a block size of 2 using a balanced design using computer-executed software. The primary endpoint is the fasting and postprandial blood glucose, insulin, and continuous glucose monitoring after fasting. Secondary endpoints include postprandial blood lipids, clock gene expressions in peripheral blood cells, and non-targeted postprandial plasma metabolome. The 2 intervention days include a no-breakfast day and a no-dinner day. The diets before, during, and after the intervention day was designed according to Dietary Guidelines for Chinese Residents (2022), and the energy distribution of three meals is 1:1:1, with the energy percentage of carbohydrate, protein, and fat being 55%, 15%, and 30%, respectively. The time of breakfast, lunch, and dinner is 7.30 a.m., 1.00 p.m., and 8.00 p.m., respectively. All participants are instructed to follow their natural dietary plans in the wash-out period, and the food intakes and sleep circle were recorded by a modified food frequency questionnaire (FFQ).

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women are eligible.
2. Age: 18-40 years old.
3. Healthy adults: no history of diabetes mellitus, no use of hypoglycemic drugs, no insulin injection.
4. All participants have a good sleep circle, with no somnipathy.

Exclusion Criteria:

1. Severe mental illness or other major medical comorbidities and autoimmune diseases (e.g., chronic renal failure, cardiovascular diseases, or cancer)
2. Skipping breakfast or dinner more than 10 times within 6 months.
3. Following a special diet, currently on weight loss medication, using sleeping medications.
4. Pregnancy or to be pregnant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from fasting to postprandial postprandial blood glucose | Blood samples collected before and after 2 hours at lunch on the no-breakfast day; blood samples collected before and after 2 hours at next day breakfast on the no-dinner day
  The primary endpoint is fasting and postprandial blood glucose with hexokinase tests.
Change from fasting to postprandial insulin | Blood samples collected before and after 2 hours at lunch on the no-breakfast day; blood samples collected before and after 2 hours at next day breakfast on the no-dinner day
  Fasting and postprandial insulin will be tested by ELISA KIT.
Results of continuous glucose monitoring | From the day before the first intervention day and the wash-out period till the day after the second intervention day (10 days in total)
  Continuous glucose will be monitored by Abott glucose monitor.

SECONDARY OUTCOMES:
Change from fasting to postprandial blood lipids | Blood samples collected before and after 2 hours at lunch on the no-breakfast day; blood samples collected before and after 2 hours at next day breakfast on the no-dinner day
  Fasting and postprandial total-, HDL-, LDL-cholesterol, triglyceride will be tested.
Analyzes of clock gene expression in peripheral blood cells (PBC) | PBC samples collected before and after 2 hours at lunch on the no-breakfast day; blood samples collected before and after 2 hours at next day breakfast on the no-dinner day
  Clock gene expression in PBC will be evaluated by RT-PCR.
Analyzes of postprandial plasma metabolome | Blood samples collected at 2 hours after each meal
  Non-targeted plasma metabolites will be tested by LC-MS-MS after 2 hours of each meal.

CONTACTS AND LOCATIONS:
Overall Officials: Yuwei Liu, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Institute of Planned Parenthood Research Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Nas A, Mirza N, Hagele F, Kahlhofer J, Keller J, Rising R, Kufer TA, Bosy-Westphal A. Impact of breakfast skipping compared with dinner skipping on regulation of energy balance and metabolic risk. Am J Clin Nutr. 2017 Jun;105(6):1351-1361. doi: 10.3945/ajcn.116.151332. Epub 2017 May 10. PMID 28490511
- [Result] Jakubowicz D, Wainstein J, Landau Z, Raz I, Ahren B, Chapnik N, Ganz T, Menaged M, Barnea M, Bar-Dayan Y, Froy O. Influences of Breakfast on Clock Gene Expression and Postprandial Glycemia in Healthy Individuals and Individuals With Diabetes: A Randomized Clinical Trial. Diabetes Care. 2017 Nov;40(11):1573-1579. doi: 10.2337/dc16-2753. Epub 2017 Aug 22. PMID 28830875
- [Result] Ogata H, Kayaba M, Tanaka Y, Yajima K, Iwayama K, Ando A, Park I, Kiyono K, Omi N, Satoh M, Tokuyama K. Effect of skipping breakfast for 6 days on energy metabolism and diurnal rhythm of blood glucose in young healthy Japanese males. Am J Clin Nutr. 2019 Jul 1;110(1):41-52. doi: 10.1093/ajcn/nqy346. PMID 31095288
- [Result] Garaulet M, Lopez-Minguez J, Dashti HS, Vetter C, Hernandez-Martinez AM, Perez-Ayala M, Baraza JC, Wang W, Florez JC, Scheer FAJL, Saxena R. Interplay of Dinner Timing and MTNR1B Type 2 Diabetes Risk Variant on Glucose Tolerance and Insulin Secretion: A Randomized Crossover Trial. Diabetes Care. 2022 Mar 1;45(3):512-519. doi: 10.2337/dc21-1314. PMID 35015083
- [Result] Lopez-Minguez J, Saxena R, Bandin C, Scheer FA, Garaulet M. Late dinner impairs glucose tolerance in MTNR1B risk allele carriers: A randomized, cross-over study. Clin Nutr. 2018 Aug;37(4):1133-1140. doi: 10.1016/j.clnu.2017.04.003. Epub 2017 Apr 10. PMID 28455106
- See also: Impact of breakfast skipping compared with dinner skipping on regulation of energy balance and metabolic risk — https://pubmed.ncbi.nlm.nih.gov/28490511/
- See also: Influences of Breakfast on Clock Gene Expression and Postprandial Glycemia in Healthy Individuals and Individuals With Diabetes: A Randomized Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/28830875/
- See also: Effect of skipping breakfast for 6 days on energy metabolism and diurnal rhythm of blood glucose in young healthy Japanese males — https://pubmed.ncbi.nlm.nih.gov/31095288/
- See also: Interplay of Dinner Timing and MTNR1B Type 2 Diabetes Risk Variant on Glucose Tolerance and Insulin Secretion: A Randomized Crossover Trial. — https://pubmed.ncbi.nlm.nih.gov/35015083/
- See also: Late dinner impairs glucose tolerance in MTNR1B risk allele carriers: A randomized, cross-over study. — https://pubmed.ncbi.nlm.nih.gov/28455106/